CLINICAL TRIAL: NCT02699580
Title: Protective Effect of Biodegradable Collagen Implant (Ologen) in Scleral Thinning After Strabismus Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 4-2015-0741
Record Dates: First submitted 2016-02-22; First posted 2016-03-04 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Exotropia or Intermittent Exotropia
Keywords: Biodegradable collagen implant; scleral thinning; strabismus surgery
MeSH Terms: conditions — Exotropia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Biodegradable collagen implant (Experimental): Both eyes are needed to correct strabismus. One eye is randomly selected for the placement of biodegradable collagen implant.
  Interventions: Device: lateral rectus recession with biodegradable collagen implant
- Without biodegradable collagen implant (Active Comparator): Strabismus surgery is done without placing of biodegradable collagen implant in the other eye.
  Interventions: Procedure: Lateral rectus recession without biodegradable collagen implantation

INTERVENTIONS:
Device: lateral rectus recession with biodegradable collagen implant — Exotropia was treated with bilateral lateral rectus recession procedure. Lateral rectus recession was done. After lateral rectus recession, no degradable collagen implant was placed in the area, where lateral rectus was original inserted. One eye was randomly selected for the comparison.
  Arms: Biodegradable collagen implant
Procedure: Lateral rectus recession without biodegradable collagen implantation — Exotropia was treated with bilateral lateral rectus recession procedure. Lateral rectus recession was done in the other eye without placing biodegradable collagen implantation.
  Arms: Without biodegradable collagen implant

SUMMARY:
This study is to investigate protective effect of biodegradable collagen implant in scleral showing after lateral rectus recession in patients with exotropia.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with intermittent exotropia or constant exotropia
2. Alternate prism cover test showed 20 prism diopters or more than 20 prism diopters exotropia
3. Subjects who want to do strabismus surgery

Exclusion Criteria:

1. Subject who had previous strabismus surgery or other ocular surgery history
2. Thyroid eye disease or other connective tissue disease
3. Significant bleeding or scleral perforation during operation
4. Subjects who need to do medial rectus resection, not lateral rectus recession
5. Subjects who had a plan to do other intra or extraocular surgery within 3 months

Ages: 10 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-09-30 (Actual); Primary Completion 2016-09-10 (Actual); Study Completion 2016-09-10 (Actual)

PRIMARY OUTCOMES:
Scleral thinning assessed with slit photography | Postoperative 3 months
  Scleral thinning at the area, where lateral rectus was originally inserted, was assessed with slit photography. Scleral thinning score was calculated from the Lab color model.

SECONDARY OUTCOMES:
Ocular discharge assessed by questionnaire | Postoperative 1 week
  Ocular discharge will be assessed by questionnaire.
Tearing assessed by questionnaire | Postoperative 1 week
  Tearing will be assessed by questionnaire.
Foreign body sensation assessed by questionnaire | Postoperative 1 week
  Foreign body sensation will be assessed by questionnaire.
Collagen implant protrusion assessed by questionnaire | Postoperative 1 week
  Collagen implant protrusion will be assessed by questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Ophthalmology, Severance Hospital, Yonsei University College of Medicine, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
no plan to share individual participant data

REFERENCES:
- [Derived] Pang Y, Gnanaraj L, Gayleard J, Han G, Hatt SR. Interventions for intermittent exotropia. Cochrane Database Syst Rev. 2021 Sep 13;9(9):CD003737. doi: 10.1002/14651858.CD003737.pub4. PMID 34516656